CLINICAL TRIAL: NCT04357613
Title: A RANDOMIZED NON-COMPARATIVE PHASE 2 PILOT STUDY TESTING THE VALUE OF IMATINIB MESYLATE AS AN EARLY TREATMENT OF COVID-19 DISEASE IN AGED HOSPITALIZED PATIENTS.
Brief Title: IMATINIB IN COVID-19 DISEASE IN AGED PATIENTS.
Acronym: IMAGE-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Philippe ROUSSELOT, MD, Versailles Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P20/05_IMAGE19
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: SARS Virus
MeSH Terms: conditions — Severe Acute Respiratory Syndrome | interventions — Drugs, Investigational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expérimental ARM (Experimental): 800mg/d IMATINIB during 14days
  Interventions: Drug: Experimental drug
- Comparator ARM (No Intervention): Standard of care

INTERVENTIONS:
Drug: Experimental drug — Imatinib 800mg/d during 14days
  Arms: Expérimental ARM

SUMMARY:
High-throughput screening studies identified Abl kinase inhibitors (including imatinib) as inhibitors of coronaviruses SARS and MERS. The SARS-CoV-2 coronavirus depend on Abl2 kinase activity to fuse and enter into the cells. Pharmacokinetic studies demonstrated that IC50 of imatinib for ABL1, BCR-ABL1 and ABL2 kinase inhibition is less than 1 microM (around 0.3 microM) below the expected trough plasmatic concentrations of imatinib 400 mg/day (1.7 microM). The EC50 of imatinib for the inhibition of the virus is under investigation but we now have a first estimates with EC50 close to 2.5 microM. This plasmatic concentration is achievable with imatinib 800 mg/d. We hypothesize that clinically achievable imatinib concentration will block the first round of cell to cell virus infection and therefore stop or prevent from SARS-CoV-2 infection in human. Based on our 20 years' experience of prescribing imatinib in patients, we expect that most of the adverse events and pharmacological interactions of imatinib can be anticipated and corrected. The eligible population will be aged (>70y) patients hospitalized for a non-severe COVID-19 disease for less than 7 days. Patients will be randomized 1/1 between standard of care and imatinib 800 mg per day during 14 days. The primary endpoint will be the death rate by 30 days. Secondary endpoint will include progression to severe CIVID-19 disease, safety, outcome at 3 months. We plan to randomize 90 patients in order to show a 10% benefit in term of death rate reduction from 16% to 6%.

ELIGIBILITY:
Inclusion Criteria:. Patient aged > 70y 2. Patient with a documented COVID-19 disease by SARS-CoV-2 RT-PCR (if no test is available, suspected COVID-19 disease on CT SCAN).

3. Initial phase (≤ 7 days) of COVID-19 disease 4. Non severe COVID-19 disease 5. Signed informe consent

Exclusion Criteria:

1. Patient in palliative care
2. Severe COVID-19 disease (SpO2 ≤ 94% with O2 ≥ 5 l/min)
3. Contra-indication to imatinib
4. Therapy with Warfarin (Heparin allowed)
5. Stage II to IV congestive heart failure (CHF) as determined by the New York Heart Association (NYHA)
6. Peripheral edema grade > 2
7. Known HBV, HBC or HIV infection
8. Known hepatic failure
9. Patient under legal protection

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the benefit of early imatinib therapy to prevent severe COVID-19 disease in hospitalized aged patients. | 30 days
  To evaluate the 30 days mortality rate in aged patients hospitalized with COVID-19

SECONDARY OUTCOMES:
To evaluate the feasibility of imatinib therapy. | Day 14
  Drop out rate of imatinib mesylate therapy
To evaluate safety of imatinib therapy | 3 months
  Adverse events related to imatinib mesylate therapy
To evaluate the clinical evolution | 3 months
  Clinical (WHO COVID scale) and geriatric scores (GIR, ADL and IADL) modification
To evaluate the progression rate to severe COVID-19 disease | 3 months
  Clinical (WHO COVID scale) and geriatric scores (GIR, ADL and IADL) modification
To evaluate mortality | 14 days
  number of death
To evaluate mortality | 60 days
  number of death
To evaluate mortality | 90 days
  number of death
To evaluate viral load | 14 days
  Viral load by SARS-CoV-2 PCR
To evaluate plasmatic levels of imatinib | 14 days
  Imatinib trough level

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Rousselot, Principal Investigator — CH Versailles
Locations (2):
- France (2):
  - CHU Bordeaux, Bordeaux
  - CH de Versailles, Le Chesnay

REFERENCES:
- [Derived] Zhao H, Mendenhall M, Deininger MW. Imatinib is not a potent anti-SARS-CoV-2 drug. Leukemia. 2020 Nov;34(11):3085-3087. doi: 10.1038/s41375-020-01045-9. Epub 2020 Sep 30. No abstract available. PMID 32999432